CLINICAL TRIAL: NCT01783353
Title: Oral Zinc Gluconate as Treatment for Recalcitrant Cutaneous Warts: A Randomized, Double-blind, Placebo-controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Philippine Dermatological Society (Network)
Responsible Party: Principal Investigator, Rochelle L. Castillo, M.D., Philippine Dermatological Society
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDS_PGH_2013_001
Record Dates: First submitted 2013-01-30; First posted 2013-02-04 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Recalcitrant Cutaneous Warts
Keywords: Recalcitrant cutaneous warts; verruca
MeSH Terms: conditions — Warts | interventions — gluconic acid; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corn starch pill (Placebo Comparator): Two (2) corn starch pills will be taken three (3) times a day for 60 days.
  Interventions: Dietary Supplement: Corn starch pill
- Zinc gluconate (Experimental): Two (2) zinc gluconate 50 mg capsules will be taken three (3) times a day for 60 days.
  Interventions: Dietary Supplement: Zinc gluconate

INTERVENTIONS:
Dietary Supplement: Zinc gluconate
  Arms: Zinc gluconate
Dietary Supplement: Corn starch pill
  Arms: Corn starch pill

SUMMARY:
Up to one-third of common warts can remain recalcitrant, an occurrence that has been attributed to impaired cell-mediated immunity. At present, no guidelines exist for the management of recalcitrant cutaneous warts. Zinc, a well-established immunomodulatory agent, has shown promise in this regard. Previous studies documenting the efficacy of oral zinc used zinc sulfate given at a maximum dose of 600 mg/day, equivalent to 140 mg of elemental zinc, which is over three times the recommended upper limit of 40 mg of elemental zinc per day. This raises concerns over safety and tolerability. In the Philippines, oral zinc is more widely available in chelated forms such as zinc gluconate, which have the benefit of improved absorption compared to non-chelated compounds such as zinc sulfate. This study will seek to determine if zinc gluconate 300 mg/day, equivalent to 40 mg of elemental zinc, will be efficacious in treating recalcitrant cutaneous warts. This lowered dose may have the added benefits of increased safety, tolerability, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female
2. Age 19 years and older
3. With ≥ one (1) recalcitrant common, mosaic, palmar, plantar, or periungual wart/s
4. Consent given

Exclusion Criteria:

1. Current or history of mental illness
2. Current or history of malignancy
3. Severe immunodeficiency states
4. Pregnant or lactating
5. Documented adverse effects to oral or topical zinc exposure
6. Oral intake of zinc supplements in the past 12 months or less
7. Oral Intake of H2 antagonists in the past 4 weeks or less
8. Oral intake of immunosuppressives in the past 4 weeks or less
9. Concurrent usage of other treatment modalities
10. Current anogenital warts

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Efficacy based on the resolution rate (i.e. the percentage of baseline warts that resolve completely) on Days 30 and 60 | 60 days

SECONDARY OUTCOMES:
Types of adverse events | 60 days
  Types and severity of adverse events will be noted on Day 30 (+5 days) and Day 60 (+5 days) by the primary investigator by verbally asking the subjects and by physically examining them
Severity of adverse events | 60 days
  Types and severity of adverse events will be noted on Day 30 (+5 days) and Day 60 (+5 days) by the primary investigator by verbally asking the subjects and by physically examining them. Severity will be based on the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events by the National Institute Of Allergy And Infectious Diseases. For abnormalities not found in the DAIDS Toxicity Tables, the following scale will be used to estimate grade:
  * Grade 1, Mild: No limitation in activity; no medical intervention/therapy required
  * Grade 2, Moderate: Mild to moderate limitation in activity; no or minimal medical intervention required
  * Grade 3, Severe: Marked limitation in activity; medical intervention required; hospitalization possible
  * Grade 4, Life-Threatening: Extreme limitation in activity; significant medical intervention required; hospitalization or hospice care probable
Recurrence | 120 days
  The recurrence rate in patients who achieve complete response to zinc will be assessed at Day 120 or two months after discontinuation of zinc intake.

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle L. Castillo, M.D., Principal Investigator — Philippine General Hospital Section of Dermatology
Locations (1):
- Philippine General Hospital, Manila, NCR, Philippines